CLINICAL TRIAL: NCT04007536
Title: A Prospective, Longitudinal Study of Potential Treatment-Responsive Biomarkers and Clinical Outcomes in Hunter Syndrome
Brief Title: A Study of Potential Treatment-Responsive Biomarkers and Clinical Outcomes in Hunter Syndrome
Status: Completed | Type: Observational
Sponsor: Denali Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DNLI-E-0001
Record Dates: First submitted 2019-06-22; First posted 2019-07-05 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Mucopolysaccharidosis II
Keywords: MPS-II; Hunter Syndrome; Lysosomal Storage Disease; nMPS II; nnMPS II
MeSH Terms: conditions — Mucopolysaccharidosis II; Sudden Infant Death; Lysosomal Storage Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, cerebrospinal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Part 1: Participants from 2 through 10 years of age who have MPS II. Clinical, neurocognitive, laboratory, and biomarker assessments will be conducted.
  Interventions: Other: No Intervention
- Part 2: Participants from 2 through 30 years of age who have MPS II; Part 2 will entail a single collection of cerebrospinal fluid (CSF), urine, and blood. Clinical outcome assessments are optional in Part 2 for participants aged 18 years or younger; no clinical assessments are planned for participants older than 18 years.
  Interventions: Other: No Intervention
- Part 3: Participants <8 years of age who have the neuronopathic form of mucopolysaccharidosis type II (nMPS II). Clinical, neurocognitive, laboratory, and biomarker assessments will be conducted.
  Interventions: Other: No Intervention
- Part 4: Participants 6 to 17 years of age with the non-neuronopathic form of mucopolysaccharidosis type II (nnMPS II). Clinical, neurocognitive, laboratory, and biomarker assessments will be conducted.
  Interventions: Other: No Intervention
- Part 5: Participants ≤3 years of age with an undetermined MPS II phenotype. Clinical, neurocognitive, laboratory, and biomarker assessments will be conducted.
  Interventions: Other: No Intervention
- Part 6: Participants from 1 to 17 years of age with nMPS II. Clinical, neurocognitive, laboratory, and biomarker assessments will be conducted. Part 6 will also include a single collection of CSF.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
This is a six-part prospective, multicenter, multiregional observational study of patients with mucopolysaccharidosis type II (MPS II), also known as Hunter syndrome, to assess biomarkers potentially related to disease severity and/or treatment response and prospectively assess the progression of disease in participants with MPS II who are aged ≤30 years at the time of enrollment.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria (Part 1):

* Participants aged 2 through 10 years
* nMPS II subgroup: participants with a development quotient (DQ) <85 and/or a decline of at least 7.5 points in DQ, assessed at least 6 months apart, or with the same genetic mutation as a blood relative with confirmed nMPS II

Key Inclusion Criteria (Part 2):

* Participants aged 2 through 30 years
* nMPS II subgroup: patients with an age-adjusted DQ <85 and/or a decline of 10 points or more in DQ in the previous 6 months or more, or with the same genetic mutation as a blood relative with confirmed nMPS II
* Scheduled to undergo general anesthesia or CSF sampling for non-study-related medical reasons and parent(s)/legally authorized representative consent to donate CSF for research purposes during that procedure, or an adult patient is able to provide consent and agrees to participation in the study for CSF collection/donation

Key Inclusion Criteria (Part 3):

* nMPS II participants aged <8 years

Key Inclusion Criteria (Part 4):

* nnMPS II participants aged 6 to 17 years

Key Inclusion Criteria (Part 5):

* Participants aged ≤ 3 years
* Have undetermined MPS II phenotype

  * Do not have a large deletion(s) or rearrangement(s) in the IDS gene or other definitive mutation indicative of nMPS II
  * Do not have a DQ < 85 at the screening/baseline neurocognitive assessment and/or a documented decline of at least 7.5 points in DQ in the previous 6 to 18 months
  * Do not have the same IDS gene variant as a blood relative with confirmed nMPS II or nnMPS II

Key Inclusion Criteria (Part 6):

* nMPS II participants aged 1 to 17 years
* Have received an MPS II gene therapy or allogeneic HSCT > 12 months prior to screening
* Have a post-HSCT or post-gene therapy DQ < 85 at the screening/baseline neurocognitive assessment and/or a documented decline of at least 7.5 points in DQ in the previous 6 to 18 months

Key Exclusion Criteria (All Parts):

* Have unstable medical condition that would make participation in the study unsafe or would interfere with necessary medical care
* Have received any central nervous system (CNS)-targeted MPS II investigational therapy within the previous 6 months

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients ≤ 30 years with a confirmed diagnosis of MPS II based on IDS (iduronate 2-sulfatase) enzyme activity and documented mutation in the IDS gene
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Changes in adaptive behavior over time as measured by Vineland Adaptive Behavior Scales, Second Edition (VABS II) and/or Vineland Adaptive Behavior Scales, Third Edition (Vineland-3) | Up to 96 weeks
Changes in neurocognition over time as measured by Bayley Scales of Infant and Toddler Development, 3rd Edition; Kaufman Assessment Battery for Children, 2nd Edition; or Wechsler Intelligence Scale for Children, Fifth Edition | Up to 96 weeks
Changes in levels of total urine glycosaminoglycans (GAGs), levels of heparan sulfate (HS) and dermatan sulfate (DS) in cerebrospinal fluid (CSF), urine and/or blood | up to 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Katia Meirelles, MD, Study Director — Denali Therapeutics
Locations (6):
- United States (3):
  - UCSF Benioff Children's Hospital, Oakland, California
  - UNC Children's Research Institute, Chapel Hill, North Carolina
  - UPMC | Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands
- United Kingdom (2):
  - Birmingham Children's Hospital, Birmingham
  - Manchester Centre for Genomic Medicine, Manchester

IPD SHARING:
Plan to Share IPD: No